CLINICAL TRIAL: NCT03260673
Title: 白内障超声乳化术对2型糖尿病患者角膜内皮细胞的影响 Corneal Endothelial Cell Changes After Phacoemulsification in Patients With Type 2 Diabetes Mellitus
Brief Title: Corneal Endothelial Cell Changes After Phacoemulsification in Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 17102
Record Dates: First submitted 2017-07-27; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Cataract; Diabetes Mellitus
Keywords: cataract; phacoemulsification; type 2 diabetes mellitus; corneal endothelial cells
MeSH Terms: conditions — Cataract; Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the diabetic group: patients with type 2 diabetes scheduled to undergo cataract surgery
  Interventions: Other: specular microscope
- the control group: patients without diabetes scheduled to undergo cataract surgery
  Interventions: Other: specular microscope

INTERVENTIONS:
Other: specular microscope — The corneal endothelial cell density, variation in endothelial cell size (CV), percentage of hexagonal cells, and central corneal thickness(CCT) were recorded at baseline and at 3 months postoperatively.

SUMMARY:
This study investigate the change of the corneal endothelial cells in patients with type 2 diabetes after phacoemulsification with intraocular lens implantation.

DETAILED DESCRIPTION:
The investigators do the clinical prospective study including 30 patients with type 2 diabetes and 30 control patients without diabetes scheduled to undergo cataract surgery. The corneal endothelial cell density, variation in endothelial cell size (CV), percentage of hexagonal cells, and central corneal thickness(CCT) were recorded at baseline and at 3 months postoperatively.Then, the investigators compared the two sets of data. At last observing the change of the corneal endothelial cells in patients with type 2 diabetes after phacoemulsification with intraocular lens implantation.

ELIGIBILITY:
Inclusion Criteria:

the experimental group:

1. Clinical diagnosis of cataract
2. Type 2 diabetes mellitus
3. The recent blood glucose control was stable
4. The glycosylated hemoglobin < 8%

The control group:

1. Clinical diagnosis of cataract
2. No history of type 2 diabetes

Exclusion Criteria:

1. Corneal lesions
2. Anterior inflammation
3. Ocular trauma or surgical history
4. Glaucoma
5. Corneal endothelial cell density < 1500 / mm squared

Ages: 58 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among the 60 patients enrolled in this study, the experimental group was 77.5 ±9.2 years old, and the control age was 76.3±8.7 years, with no statistical difference (P = 0.87). All patients were treated for 3 months.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Comparison of the corneal endothelial cell density before-after cataract surgery | half year
  Comparison of the corneal endothelial cell density before-after cataract surgery，the density is expressed in terms of the number of cells per square millimeter.

SECONDARY OUTCOMES:
Comparison of the endothelial cell size before-after cataract surgery | half year
  Comparison of the endothelial cell size before-after cataract surgery，the size is measured in square microns.
Comparison of the percentage of hexagonal cells before-after cataract surgery | half year
  Comparison of the percentage of hexagonal cells before-after cataract surgery,the percentage are expressed as "%".
Comparison of the central corneal thickness(CCT) before-after cataract surgery | half year
  Comparison of the central corneal thickness(CCT) before-after cataract surgery，the thickness is in microns.

IPD SHARING:
Plan to Share IPD: Yes